CLINICAL TRIAL: NCT07355504
Title: Prostate Cancer Early Detection Using Serial MRI Examinations
Acronym: PROCEDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC24.0296
Record Dates: First submitted 2025-12-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: MRI lesion
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate biopsy (No Intervention): Patients randomized to the standard of care arm will undergo prostate biopsies
- MRI surveillance (Experimental): Patients randomized to the experimental arm will proceed with MRI surveillance.
  Interventions: Procedure: MRI Examination

INTERVENTIONS:
Procedure: MRI Examination — Patients randomized to the experimental arm will proceed with MRI surveillance. A follow-up visit is planned at 6 months with the result of a PSA test, and it is possible at each investigator's discretion, to prescribe the follow-up MRI at 6 months in case of rising PSA. Otherwise, the repeat MRI will be scheduled one year after the initial MRI. Images will also be sent to the coordinating center for central reviewing of the new MRI exam and assessment of progression.
  Arms: MRI surveillance

SUMMARY:
The rationale of the PROCEDE trial is to explore a novel early detection strategy in which biopsy decision does not rely on one single MRI examination, but on the progression of the MRI lesion between 2 consecutive exams, with the objective of reducing the number of unnecessary biopsies, detection of non-clinically prostate cancer and, ultimately, overtreatment.

ELIGIBILITY:
Inclusion Criteria:

* Men aged over 18 years
* Men with an estimated life expectancy of more than 10 years
* Biopsy-naïve men
* PSA level ≤ 20 ng/ml
* Presence, on the first multiparametric prostate MRI, of a PIRADS 3-5 lesion confirmed by local rereading if the MRI was performed outside the center
* MRI of sufficient quality (PI-QUAL score 2-3)
* PIRADS 3 lesion with a PSA density <0.15 ng/ml/ml
* No signs of extracapsular extension or seminal vesicle invasion (MRI stage T2 confirmed by local rereading if MRI performed outside the center)
* No suspicious lymph node (confirmed by local rereading if MRI performed outside the center)
* Patient is insured (affiliated with the national health insurance system or benefiting from such coverage)
* Signed informed consent form

Exclusion Criteria:

* Men already under surveillance for a known MRI lesion (except if the previous MRI was performed less than 6 months ago)
* Known mutation in DNA repair genes or suggestive family history
* PIRADS 3 lesion with PSA density < 0.15 ng/ml/ml
* PIRADS 5 lesion with suspected extracapsular extension or seminal vesicle invasion
* Suspicion of lymph node involvement
* Multiparametric prostate MRI showing a PIRADS 1-2 lesion
* Use of treatments that may modify the appearance of MRI lesions: 5-alpha reductase inhibitors, hormone therapy
* Patient with severe renal insufficiency (GFR < 30 ml/min/1.73 m²)
* Contraindication to gadolinium injection
* Contraindication to prostate biopsy
* Vulnerable persons (covered by Articles L1111-6 to L1111-8 of the French Public Health Code)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-01-24 (Estimated); Study Completion 2033-01-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of a novel early detection strategy based on serial MRI | at 2 years
  To evaluate the impact of a novel early detection strategy based on serial MRI exams, compared to the standard of care, on the rate of definitive treatment for localized prostate cancer

SECONDARY OUTCOMES:
To assess the impact of a new early-detection strategy based on repeated MRI | at 5 years.
  Time to the first event among (i) definitive treatment for localized prostate cancer, defined as one of the following procedures: radical prostatectomy, radiotherapy, brachytherapy, focal therapy; (ii) occurrence of prostate cancer metastases; (iii) all-cause death, occurring between randomization and 5-year follow-up.
To assess the impact of the new strategy on the number of prostate biopsies performed | at 2 years and 5 years.
  Number of biopsy procedures performed.
To assess changes in therapeutic options with the new strategy | at 2 years and 5 years.
  Choice of definitive treatment, if applicable, among the following options: (i) brachytherapy, (ii) focal therapy, and (iii) unimodal therapy.
To assess the oncologic safety with Adverse pathological criteria (pT3, pN1, detectable PSA)of the new strategy compared with the usual strategy | at 2 years and 5 years.
  Adverse pathological criteria (pT3, pN1, detectable PSA) in patients treated with radical prostatectomy.
To assess the oncologic outcomes (Biochemical recurrence-free survival, disease-specific survival and overall survival.of the new strategy compared with the usual strategy | at 2 years and 5 years.
  Biochemical recurrence-free survival, disease-specific survival (i.e., censoring non-disease-related deaths), and overall survival.
To assess the impact of the new strategy on patients' anxiety levels and quality of life, evaluated at Day 0 and then annually for 5 years. | at 5 years
  HADS scale, MAX-PC questionnaire, EPIC-26 questionnaire, EQ-5D-5L questionnaire.
  The combination of these questionnaires will allow us to assess the level of anxiety and the quality of life of patients treated with the new strategy; we have decided to use them together for a combined evaluation.
To evaluate the cost-effectiveness of the new early-detection strategy compared with the standard of care from a societal perspective | at 5 years.
  ICUR. The incremental cost-utility ratio (ICUR) will be calculated by dividing the mean difference in costs by the mean difference in QALYs (estimated from the EQ-5D-5L). The ratio will be expressed as cost per healthy life-year gained.
To establish an MRI database enabling comparison of radiomic characteristics between patients who have progressed and those who have not, in order to identify new imaging features associated with disease progression. | at 5 years
  Database collecting all MRI examinations in DICOM format, along with oncologic outcomes (progression/no progression).

CONTACTS AND LOCATIONS:
Locations (1):
- university Hospital Grenoble, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No